CLINICAL TRIAL: NCT01607892
Title: A Phase I Study of the Safety, Pharmacokinetics and Pharmacodynamics of Escalating Doses of the Selective Inhibitor of Nuclear Export/SINE™ Compound KPT-330 in Patients With Advanced Hematological Malignancies
Brief Title: Safety Study of the Selective Inhibitor of Nuclear Export (SINE) KPT-330 in Patients With Advanced Hematological Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-001
Record Dates: First submitted 2012-05-16; First posted 2012-05-30 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Hematological Malignancies
Keywords: Selinexor; KPT-330; Multiple Myeloma; non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Waldenström's macroglobulinemia; Peripheral T-Cell Lymphoma; Cutaneous T-Cell Lymphoma; Chronic Myelocytic Leukemia; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- selinexor (Experimental)
  Interventions: Drug: KPT-330

INTERVENTIONS:
Drug: KPT-330
  Other Names: Selinexor

SUMMARY:
The purpose of this research study is to find out more information relating to the highest dose of KCP-330 that can be given safely and side effects it may cause, to examine how the body affects KCP-330 concentrations in the blood (pharmacokinetics or PK), to examine the effects of KCP-330 on the body (pharmacodynamics or PDn) and to obtain information on its effectiveness in treating cancer.

ELIGIBILITY:
Inclusion Criteria

1. Malignancies that are refractory to or intolerant of established therapy known to provide clinical benefit. Patients must not be candidates for anti-tumor regimes known to provide clinical benefit.
2. All patients must have evidence of progressive disease on study entry. Previously untreated patients who are not chemotherapy candidates on Arm 2 may have advanced disease (without clear progression). There is no upper limit on the number of prior treatments provided that all inclusion criteria are met, and exclusion criteria are not met.

Exclusion Criteria

1. Radiation, chemotherapy, or immunotherapy or any other anticancer therapy ≤2 weeks prior to cycle 1 day 1 and mitomycin C and radioimmunotherapy 6 weeks prior to cycle 1 day 1.
2. Patients with active graft versus host disease after allogeneic stem cell transplantation. At least 3 months must have elapsed since completion of allogeneic stem cell transplantation except for patients with AML, where at least 2 months must have elapsed;
3. Known active hepatitis A, B, or C infection; or known to be positive for HCV RNA or HBsAg (HBV surface antigen);
4. Patients with active CNS malignancy. Asymptomatic small lesions are not considered active. Treated lesions may be considered inactive if they are stable for at least 3 months. Patient with malignant cells in their cerebrospinal fluid (CSF) without CNS symptom may be included.
5. Significantly diseased or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea.
6. Grade ≥2 peripheral neuropathy at baseline (within 14 days prior to cycle 1 day 1).
7. Macular degeneration, uncontrolled glaucoma, or markedly decreased visual acuity.
8. In the opinion of the investigator, patients who are significantly below their ideal body weight.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2012-07-23 (Actual); Primary Completion 2015-10-13 (Actual); Study Completion 2015-10-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (9):
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical Center, New York, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - The Ohio State University, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Princess Margaret Hospital, Toronto, Ontario
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chen C, Siegel D, Gutierrez M, Jacoby M, Hofmeister CC, Gabrail N, Baz R, Mau-Sorensen M, Berdeja JG, Savona M, Savoie L, Trudel S, Areethamsirikul N, Unger TJ, Rashal T, Hanke T, Kauffman M, Shacham S, Reece D. Safety and efficacy of selinexor in relapsed or refractory multiple myeloma and Waldenstrom macroglobulinemia. Blood. 2018 Feb 22;131(8):855-863. doi: 10.1182/blood-2017-08-797886. Epub 2017 Dec 4. PMID 29203585
- [Derived] Kuruvilla J, Savona M, Baz R, Mau-Sorensen PM, Gabrail N, Garzon R, Stone R, Wang M, Savoie L, Martin P, Flinn I, Jacoby M, Unger TJ, Saint-Martin JR, Rashal T, Friedlander S, Carlson R, Kauffman M, Shacham S, Gutierrez M. Selective inhibition of nuclear export with selinexor in patients with non-Hodgkin lymphoma. Blood. 2017 Jun 15;129(24):3175-3183. doi: 10.1182/blood-2016-11-750174. Epub 2017 May 3. PMID 28468797
- [Derived] Garzon R, Savona M, Baz R, Andreeff M, Gabrail N, Gutierrez M, Savoie L, Mau-Sorensen PM, Wagner-Johnston N, Yee K, Unger TJ, Saint-Martin JR, Carlson R, Rashal T, Kashyap T, Klebanov B, Shacham S, Kauffman M, Stone R. A phase 1 clinical trial of single-agent selinexor in acute myeloid leukemia. Blood. 2017 Jun 15;129(24):3165-3174. doi: 10.1182/blood-2016-11-750158. Epub 2017 Mar 23. PMID 28336527
- [Derived] Schmidt J, Braggio E, Kortuem KM, Egan JB, Zhu YX, Xin CS, Tiedemann RE, Palmer SE, Garbitt VM, McCauley D, Kauffman M, Shacham S, Chesi M, Bergsagel PL, Stewart AK. Genome-wide studies in multiple myeloma identify XPO1/CRM1 as a critical target validated using the selective nuclear export inhibitor KPT-276. Leukemia. 2013 Dec;27(12):2357-65. doi: 10.1038/leu.2013.172. Epub 2013 Jun 11. PMID 23752175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 sites in United States, Canada and Europe between 23 July 2012 (first participant treated) and 13 October 2015 (last participant completed).
Pre-assignment Details: A total of 286 participants were enrolled out of which 1 participants with MM never treated due to disease progression prior to dose initiation and 285 participants received treatment in 11 different schedules. The schedules were either 28 days (Schedules 1-7, 9-11) or 21 days (Schedule 8) per cycle and participants were treated once weekly (Schedule 7), twice weekly (Schedules 3-6, 8-11) or three times weekly alternating with 2 times weekly (Schedules 1, 2).
Groups:
- Diffuse Large B-cell Lymphoma (DLBCL): Participants with DLBCL received Selinexor in different Schedules; Schedule 1: <= 12 milligram per square meter (mg/m^2) per orally (PO) alternating 3 times per week with twice weekly dosing (1 day between doses); Schedule 2: > 12 mg/m^2 PO 3 times weekly for Week -1 followed by same dosing frequency as schedule 1 for Weeks 1-4; Schedule 3: >=30 mg/m^2 PO twice weekly (1 day between doses); Schedule 4: >=23 mg/m^2 PO twice weekly (0 days between doses) to evaluate consecutive dosing; Schedule 5: >=30 mg/m^2 PO twice weekly (2 days between doses) to evaluate dosing 2 days apart vs. 1 day apart (Schedule 3); Schedule 8: >=40 mg/m^2 PO twice weekly (1 day between doses) during Weeks 1 and 2; Schedule 9: >=45 mg/m^2 PO twice weekly in combination with 375 mg/m^2 dose of rituximab intravenous (IV) once weekly for Weeks 1-4 during different cycles. Each cycle was of 28 days (Schedule 8: 21 days of cycle) or 10 scheduled selinexor doses.
- Non-Hodgkin Lymphoma (NHL) Excluding DLBCL: Participants with NHL received Selinexor in different Schedules; Schedule 1: <= 12 mg/m^2 PO alternating 3 times per week with twice weekly dosing (1 day between doses); Schedule 2: > 12 mg/m^2 PO 3 times weekly for week -1 followed by same dosing frequency as schedule 1 for Weeks 1-4; Schedule 3: >=30 mg/m^2 PO twice weekly (1 day between doses); Schedule 5: >=30 mg/m^2 PO twice weekly (2 days between doses) to evaluate dosing 2 days apart vs 1 day apart (Schedule 3); Schedule 7: >=45 mg/m^2 PO once weekly (6 days between doses) to evaluate vs twice weekly (Schedules 3, 4, 5, and 6); Schedule 8: >=40 mg/m^2 PO twice weekly [1 Day between doses] during weeks 1 and 2; Schedule 9: >=45 mg/m^2 PO twice weekly in combination with 375 mg/m^2 dose of rituximab IV once weekly for Weeks 1-4) during different cycles. Each cycle was of 28 days (Schedule 8: 21 days of cycle) or 10 scheduled selinexor doses.
- Multiple Myeloma (MM): Participants with MM received Selinexor in different Schedules; Schedule 1: <= 12 mg/m^2 PO alternating 3 times per week with twice weekly dosing (1 Day between doses); Schedule 2: > 12 mg/m^2 3 times weekly for Week -1 followed by same dosing frequency as schedule 1 for Weeks 1-4; 3 doses (36 mg/m^2 total) in the 1-week run-in period; Schedule 3: >=30 mg/m^2 PO twice weekly (1 day between doses); Schedule 4: >=23 mg/m^2 PO twice weekly (0 days between doses) to evaluate consecutive dosing; Schedule 5: >=30 mg/m^2 PO twice weekly (2 days between doses) to evaluate dosing 2 days apart vs. 1 day apart (Schedule 3); Schedule 6: >= 35 mg/m^2 PO twice weekly with dexamethasone (20 mg twice weekly) on Days of twice weekly Selinexor dosing; Schedule 11: Group A: 40 mg; Group B: 60 mg; Group C: 80 mg twice weekly (Weeks 1, 2, and 3) at 3 fixed dose levels during different cycles. Each cycle was of 28 days or 10 scheduled selinexor doses.
- Acute Myeloid Leukemia (AML): Participants with AML received Selinexor in different Schedules; Schedule 2: > 12 mg/m^2 3 times weekly for Week -1 followed by same dosing frequency as schedule 1 for Weeks 1-4; Schedule 3: >=30 mg/m^2 PO twice weekly (1 day between doses); Schedule 5: >=30 mg/m^2 PO twice weekly (2 days between doses) to evaluate dosing 2 days apart vs. 1 day apart (Schedule 3), Schedule 7: >=45 mg/m^2 PO once weekly (6 Days between doses) to evaluate vs. twice weekly (Schedules 3, 4, 5, and 6); Schedule 8: >=40 mg/m^2 PO twice weekly (1 Day between doses) during Weeks 1 and 2; Schedule 10: >= 55 mg/m^2 PO twice weekly PO (Weeks 1 and 2) in participants with AML/18-Day treatment-free interval) during different cycles. Each cycle was of 28 days (for schedule 8: 21-day of cycle) or 10 scheduled selinexor doses.
- Other Hematological Malignancies (ALL, CML and CLL): Participants with other hematological malignancies (Acute lymphoblastic leukemia [ALL], Chronic myelogenous leukemia [CML] and chronic lymphocytic leukemia [CLL]) received Schedule 2: > 12 mg/m^2 3 times weekly for Week -1 followed by same dosing frequency as schedule 1 for Weeks 1-4; Schedule 3: >=30 mg/m^2 PO twice weekly [1 day between doses]; Schedule 4: >=23 mg/m^2 PO twice weekly (0 days between doses) to evaluate consecutive dosing; Schedule 5: >=30 mg/m^2 PO twice weekly (2 days between doses) to evaluate dosing 2 days apart vs. 1 day apart (Schedule 3); Schedule 7: >=45 mg/m^2 PO once weekly (6 Days between doses) to evaluate vs. twice weekly (Schedules 3, 4, 5, and 6); Schedule 9: >=45 mg/m^2 PO twice weekly in combination with 375 mg/m^2 dose of rituximab IV once weekly for Weeks 1-4 during different cycles. Each cycle was of 28 days or 10 scheduled selinexor doses.
Period: Overall Study
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Non-Hodgkin Lymphoma (NHL) Excluding DLBCL | Multiple Myeloma (MM) | Acute Myeloid Leukemia (AML) | Other Hematological Malignancies (ALL, CML and CLL)
Started | 58 | 27 | 81 | 95 | 24
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 58 | 27 | 81 | 95 | 24
Not completed — Need of treatment not allowed per protocol | 0 | 0 | 0 | 1 | 0
Not completed — Death | 4 | 2 | 8 | 10 | 3
Not completed — Investigator discretion | 2 | 4 | 4 | 8 | 0
Not completed — Other treatments became available | 1 | 1 | 0 | 0 | 2
Not completed — Intercurrent illness | 1 | 0 | 0 | 3 | 0
Not completed — Non-Compliance with study procedures | 0 | 0 | 1 | 0 | 0
Not completed — Consent withdrawn by participant | 9 | 4 | 24 | 14 | 4
Not completed — Disease progression | 38 | 13 | 37 | 57 | 9
Not completed — Incidence or severity of Adverse events | 3 | 3 | 7 | 2 | 6

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants who received at least 1 dose of selinexor.
Groups:
- Total: Total of all reporting groups
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Non-Hodgkin Lymphoma (NHL) Excluding DLBCL | Multiple Myeloma (MM) | Acute Myeloid Leukemia (AML) | Other Hematological Malignancies (ALL, CML and CLL) | Total
Number analyzed (Participants) | 58 | 27 | 81 | 95 | 24 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (14.00) | 58.0 (15.90) | 62.1 (8.76) | 65.6 (15.33) | 60.9 (15.23) | 61.9 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 9 | 38 | 40 | 8 | 123
  Male | 30 | 18 | 43 | 55 | 16 | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 4 | 2 | 0 | 9
  Not Hispanic or Latino | 52 | 23 | 72 | 88 | 23 | 258
  Unknown or Not Reported | 4 | 3 | 5 | 5 | 1 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 52 | 20 | 65 | 88 | 23 | 248
  Black | 2 | 3 | 11 | 5 | 1 | 22
  Asian | 0 | 1 | 4 | 1 | 1 | 7
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  American Indian or Alaskan Native | 0 | 1 | 0 | 0 | 0 | 1
  Other | 0 | 2 | 1 | 0 | 0 | 3
  Unknown/Not Reported | 4 | 0 | 0 | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product during the course of a study and which does not necessarily have to have a causal relationship with this treatment. An Serious adverse event (SAE) was an AE resulting in any of the following outcomes: death; life-threatening event; required or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. TEAEs are any untoward medical incidence in a participant during administered study treatment, whether or not these events were related to study treatment.
Time Frame: From first dose of study drug administration to end of treatment (up to 27 months)
Population: Safety population consisted of all participants who received at least 1 dose of selinexor.
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Non-Hodgkin Lymphoma (NHL) Excluding DLBCL | Multiple Myeloma (MM) | Acute Myeloid Leukemia (AML) | Other Hematological Malignancies (ALL, CML and CLL)
Number analyzed (Participants) | 58 | 27 | 81 | 95 | 24
Participants
  At Least One TEAE | 58 | 27 | 81 | 95 | 24
  At Least One Serious TEAE | 33 | 7 | 52 | 73 | 13

2. Primary Outcome: Recommended Phase 2 Dose (RP2D) of Selinexor
Description: Recommended Phase 2 dose was determined by maximum tolerated dose (MTD). MTD was defined as the next lower dose level below the one in which > 1 of 3 participants or ≥ 2 of 6 participants experienced dose-limiting toxicity (DLT), provided that that dose level is ≤25% lower than the highest dose tested. If the projected MTD was >25% lower than the highest dose tested, then an additional cohort of ≥3 participants were added at a dose that was intermediate between the intolerable dose and the next lower dose.
Time Frame: From first dose of study drug administration to end of treatment (up to 27 months)
Population: Efficacy analysis set included all participants who had either completed 1 cycle of treatment or discontinued treatment prior to completing the first cycle due to documented progressive disease (PD), death related to disease, or treatment-related toxicity. Here, data was not planned and analyzed based on individual specific disease, hence overall data was analyzed for this outcome measure.
Measure: Number; unit: milligram per square meter (mg/m^2)
Groups:
- Advanced Hematological Malignancies.: Participants received selinexor doses of <= 12 mg/m^2, post oral for all cycles 3 times weekly for Weeks 1 and 3 in schedule 1; >12 mg/m^2 3 times weekly for Weeks 2 and 4 in schedule 2; >=30 mg/m^2 on Day 1 and 3 in schedule 3; >= 23 mg/m^2 on Day 1 and Day 2 for a 28-day cycle in schedule 4; >= 30 mg/m^2 on Day 1 and 4 in schedule 5; >= 35 mg/m^2 combined with dexamethasone 20 mg on Day 1 and 3 in schedule 6; >= 45 mg/m^2 once-weekly in schedule 7; >= 40 mg/m^2 twice-weekly for first 2 weeks on Days 1, 3, 8, and 10 followed by an 11-day treatment-free interval in schedule 8; >= 30 mg/m^2 twice weekly for 3 weeks in 28-day cycle followed by fixed dose of 375 mg/m^2 Rituximab in schedule 9; 55 mg/m^2 twice-weekly on Days 1, 3, 8, and 10 followed by 18-day treatment-free interval in schedule 10; 40, 60, 80 mg (group A, group B, group C) twice weekly during the first 3 weeks, on Days 1, 3, 8, 10, 15 and 17 followed by an 11-day treatment-free interval (Days 18 through 28) in schedule 11.
Arm/Group | Advanced Hematological Malignancies.
Number analyzed (Participants) | 285
milligram per square meter (mg/m^2) | 35

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Selinexor
Description: Cmax was defined as the maximum observed concentration, taken directly from the plasma concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 24 and 48 hours post-dose on Day 1, 8 of Cycle 1 and Days 15, 16 or 17 of Cycle 2
Population: Pharmacokinetic (PK) analysis was defined as all participants who received active drug, selinexor, without the co-administration of another chemotherapeutic (i.e., rituximab), and for whom the PK profile for cycle 1 day1 (C1D1) could be adequately characterized. Here 'Overall Number of Participants Analyzed' signifies number of participants analyzed for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Selinexor (3 mg/m^2): Participants received selinexor dose of 3 mg/m^2 orally at Cycle 1, on Day 1, 3, 5, 8, 10, 15, 17, 19, 22 and 24 in schedule 1.
- Selinexor (6 mg/m^2): Participants received selinexor dose of 6 mg/m^2 orally at Cycle 1, on Day 1, 3, 5, 8, 10, 15, 17, 19, 22 and 24 in schedule 1.
- Selinexor (12 mg/m^2): Participants received selinexor dose of 12 mg/m^2 orally at Cycle 1, on Day 1, 3, 5, 8, 10, 15, 17, 19, 22 and 24 in schedule 1.
- Selinexor (16.8 mg/m^2): Participants received selinexor dose of 16.8 mg/m^2 orally at Cycle 1, on Day 1, 3, 5, 8, 15, 17, 19, and 22 in schedule 2.
- Selinexor (23 mg/m^2): Participants received selinexor dose of 23 mg/m^2 orally at Cycle 1, on Day 1 and 2 of each week for a 28-day cycle in schedule 4.
- Selinexor (30 mg/m^2): Participants received selinexor dose of 30 mg/m^2 orally at Cycle 1, on Day 1, 3, 4, 8, 10, 15 and 17 in schedule 3, 5 and 9.
- Selinexor (35 mg/m^2): Participants received selinexor dose of 35 mg/m^2 orally at Cycle 1, on Day 1 and 3 in schedule 6.
- Selinexor (40 mg/m^2): Participants received selinexor dose of 40 mg/m^2 orally at Cycle 1, on Day 1, 3, 8, 10, 15, 17 followed by an 11-day treatment-free interval (Days 18 through 28) in schedule 8 and 11.
- Selinexor (46 mg/m^2): Participants received selinexor dose of 46 mg/m^2 orally at Cycle 1, on Day 1 once-weekly in schedule 7.
- Selinexor (55 mg/m^2): Participants received selinexor dose of 55 mg/m^2 orally at Cycle 1, on Day 1, 3, 8, and 10, followed by an 18-day treatment-free interval (Days 11 through 28) in schedule 10.
- Selinexor (60 mg/m^2): Participants received selinexor dose of 60 mg/m^2 orally at Cycle 1, on Day 1, 3, 8, 10, 15, and 17, followed by an 11-day treatment-free interval (Days 18 through 28) in schedule 11.
- Selinexor (70 mg/m^2): Participants received selinexor dose of 70 mg/m^2 orally at Cycle 1, on Day 1, 3, 8, 10, 15, and 17, followed by an 11-day treatment-free interval (Days 18 through 28) in schedule 11.
- Selinexor (80 mg/m^2): Participants received selinexor dose of 80 mg/m^2 orally at Cycle 1, on Day 1, 3, 8, 10, 15, and 17, followed by an 11-day treatment-free interval (Days 18 through 28) in schedule 11.
Arm/Group | Selinexor (3 mg/m^2) | Selinexor (6 mg/m^2) | Selinexor (12 mg/m^2) | Selinexor (16.8 mg/m^2) | Selinexor (23 mg/m^2) | Selinexor (30 mg/m^2) | Selinexor (35 mg/m^2) | Selinexor (40 mg/m^2) | Selinexor (46 mg/m^2) | Selinexor (55 mg/m^2) | Selinexor (60 mg/m^2) | Selinexor (70 mg/m^2) | Selinexor (80 mg/m^2)
Number analyzed (Participants) | 2 | 3 | 6 | 13 | 18 | 21 | 13 | 8 | 9 | 8 | 4 | 8 | 5
nanogram per milliliter (ng/mL) | 49.0 (NA) — Geometric coefficient of variation (CV) was not calculated as data were available for only two participants. | 50.0 (61.1) | 149 (37.6) | 205 (46.8) | 262 (37.5) | 387 (37.1) | 407 (44.4) | 416 (36.6) | 670 (18.5) | 583 (41.4) | 668 (33.2) | 800 (32.4) | 1068 (49.3)

4. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Selinexor
Description: Tmax was defined as time of first observation of Cmax, taken directly from the plasma concentration data.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 24 and 48 hours post-dose on Day 1, 8 of Cycle 1 and Days 15, 16 or 17 of Cycle 2
Population: PK analysis was defined as all participants who received active drug, selinexor, without the co-administration of another chemotherapeutic (i.e., rituximab), and for whom the PK profile for C1D1 could be adequately characterized. Here 'Overall Number of Participants Analyzed' signifies number of participants analyzed for this outcome measure.
Measure: Median (Full Range); unit: hour
Arm/Group | Selinexor (3 mg/m^2) | Selinexor (6 mg/m^2) | Selinexor (12 mg/m^2) | Selinexor (16.8 mg/m^2) | Selinexor (23 mg/m^2) | Selinexor (30 mg/m^2) | Selinexor (35 mg/m^2) | Selinexor (40 mg/m^2) | Selinexor (46 mg/m^2) | Selinexor (55 mg/m^2) | Selinexor (60 mg/m^2) | Selinexor (70 mg/m^2) | Selinexor (80 mg/m^2)
Number analyzed (Participants) | 2 | 3 | 6 | 13 | 18 | 21 | 13 | 8 | 9 | 8 | 4 | 8 | 5
hour | NA [2.1 to 2.2] — Median value was not calculated due to insufficient PK samples required for calculation. | 4.0 [2.1 to 7.7] | 3.0 [1.1 to 4.2] | 2.08 [0.92 to 8.5] | 2.0 [1.0 to 7.8] | 2.0 [0.72 to 4.4] | 2.0 [0.92 to 4.1] | 4.0 [2.0 to 7.5] | 2.0 [0.50 to 4.2] | 2.9 [1.0 to 8.0] | 1.9 [1.8 to 2.0] | 2.0 [1.0 to 4.0] | 2.0 [0.5 to 4.0]

5. Secondary Outcome: Average Concentration From Time 0 to 24 Hours (Cavg0-24h) of Selinexor
Description: Cavg0-24h was defined as average concentration from time 0 to 24 hours.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 24 and 48 hours post-dose on Day 1, 8 of Cycle 1 and Days 15, 16 or 17 of Cycle 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Selinexor (3 mg/m^2) | Selinexor (6 mg/m^2) | Selinexor (12 mg/m^2) | Selinexor (16.8 mg/m^2) | Selinexor (23 mg/m^2) | Selinexor (30 mg/m^2) | Selinexor (35 mg/m^2) | Selinexor (40 mg/m^2) | Selinexor (46 mg/m^2) | Selinexor (55 mg/m^2) | Selinexor (60 mg/m^2) | Selinexor (70 mg/m^2) | Selinexor (80 mg/m^2)
Number analyzed (Participants) | 2 | 3 | 6 | 12 | 17 | 19 | 13 | 8 | 9 | 6 | 3 | 4 | 1
ng/mL | 17.0 (NA) — Geometric CV was not calculated as data were available for only two participants. | 20.3 (94.8) | 61.8 (39.9) | 79.0 (61.8) | 108 (46.8) | 160 (38.0) | 168 (54.0) | 163 (29.2) | 297 (26.3) | 208 (19.1) | 337 (4.2) | 353 (26.2) | NA (NA) — Geometric mean and CV were not calculated as data were available for only one participant.

6. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to t (AUC0-t) of Selinexor
Description: AUC0-t was defined as area under the concentration-time curve from time zero to the last non-zero concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 24 and 48 hours post-dose on Day 1, 8 of Cycle 1 and Days 15, 16 or 17 of Cycle 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram* hours per milliliter
Arm/Group | Selinexor (3 mg/m^2) | Selinexor (6 mg/m^2) | Selinexor (12 mg/m^2) | Selinexor (16.8 mg/m^2) | Selinexor (23 mg/m^2) | Selinexor (30 mg/m^2) | Selinexor (35 mg/m^2) | Selinexor (40 mg/m^2) | Selinexor (46 mg/m^2) | Selinexor (55 mg/m^2) | Selinexor (60 mg/m^2) | Selinexor (70 mg/m^2) | Selinexor (80 mg/m^2)
Number analyzed (Participants) | 2 | 3 | 6 | 13 | 18 | 21 | 13 | 8 | 9 | 8 | 4 | 8 | 5
nanogram* hours per milliliter | 331 (NA) — Geometric CV was not calculated as data were available for only two participants. | 564 (41.9) | 1459 (20.5) | 1829 (23.3) | 2774 (36.7) | 3461 (26.9) | 3901 (29.2) | 4481 (23.8) | 5228 (21.6) | 5601 (36.2) | 5282 (57.9) | 5466 (45.7) | 5544 (33.2)

7. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Selinexor
Description: AUC0-inf was defined as the area under the concentration-time curve from time zero to infinity (extrapolated).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 24 and 48 hours post-dose on Day 1, 8 of Cycle 1 and Days 15, 16 or 17 of Cycle 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Selinexor (3 mg/m^2) | Selinexor (6 mg/m^2) | Selinexor (12 mg/m^2) | Selinexor (16.8 mg/m^2) | Selinexor (23 mg/m^2) | Selinexor (30 mg/m^2) | Selinexor (35 mg/m^2) | Selinexor (40 mg/m^2) | Selinexor (46 mg/m^2) | Selinexor (55 mg/m^2) | Selinexor (60 mg/m^2) | Selinexor (70 mg/m^2) | Selinexor (80 mg/m^2)
Number analyzed (Participants) | 2 | 2 | 6 | 12 | 12 | 21 | 13 | 8 | 9 | 7 | 3 | 4 | 1
ng*h/mL | 348 (NA) — Geometric CV was not calculated as data were available for only two participants. | 733 (NA) — Geometric CV was not calculated as data were available for only two participants. | 1529 (18.7) | 1867 (23.6) | 2645 (1111) | 3513 (26.0) | 3948 (28.6) | 4552 (23.7) | 5284 (21.0) | 6089 (32.3) | 6964 (12.2) | 7803 (8.5) | NA (NA) — Geometric mean and CV were not calculated as data were available for only one participant.

8. Secondary Outcome: Apparent Volume of Distribution Uncorrected for Fraction Absorbed (Vd/F) of Selinexor
Description: Apparent volume of distribution was calculated as Dose/ (kel *AUC0-inf), uncorrected for fraction absorbed, reported normalized by participant body weight (kilogram [kg]).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 24 and 48 hours post-dose on Day 1, 8 of Cycle 1 and Days 15, 16 or 17 of Cycle 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per kilogram (L/kg)
Arm/Group | Selinexor (3 mg/m^2) | Selinexor (6 mg/m^2) | Selinexor (12 mg/m^2) | Selinexor (16.8 mg/m^2) | Selinexor (23 mg/m^2) | Selinexor (30 mg/m^2) | Selinexor (35 mg/m^2) | Selinexor (40 mg/m^2) | Selinexor (46 mg/m^2) | Selinexor (55 mg/m^2) | Selinexor (60 mg/m^2) | Selinexor (70 mg/m^2) | Selinexor (80 mg/m^2)
Number analyzed (Participants) | 2 | 2 | 6 | 12 | 12 | 21 | 13 | 8 | 9 | 7 | 3 | 4 | 1
Liter per kilogram (L/kg) | 1.6 (NA) — Geometric CV was not calculated as data were available for only two participants. | 1.5 (NA) — Geometric CV was not calculated as data were available for only two participants. | 1.9 (21.2) | 1.9 (29.9) | 1.9 (34.1) | 1.7 (24.1) | 2.0 (30.3) | 1.7 (29.1) | 1.8 (12.9) | 1.9 (27.9) | 1.6 (23.0) | 1.7 (13.4) | NA (NA) — Geometric mean and CV were not calculated as data were available for only one participant.

9. Secondary Outcome: Apparent Total Body Clearance, Uncorrected for Fraction Absorbed (Cl/F) of Selinexor
Description: Cl/F was calculated as Dose/AUC0-inf, uncorrected for fraction absorbed, reported normalized by participant body weight (kg).
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 24 and 48 hours post-dose on Day 1, 8 of Cycle 1 and Days 15, 16 or 17 of Cycle 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour per kilogram (L/h/kg)
Arm/Group | Selinexor (3 mg/m^2) | Selinexor (6 mg/m^2) | Selinexor (12 mg/m^2) | Selinexor (16.8 mg/m^2) | Selinexor (23 mg/m^2) | Selinexor (30 mg/m^2) | Selinexor (35 mg/m^2) | Selinexor (40 mg/m^2) | Selinexor (46 mg/m^2) | Selinexor (55 mg/m^2) | Selinexor (60 mg/m^2) | Selinexor (70 mg/m^2) | Selinexor (80 mg/m^2)
Number analyzed (Participants) | 2 | 2 | 6 | 12 | 12 | 21 | 13 | 8 | 9 | 7 | 3 | 4 | 1
Liter per hour per kilogram (L/h/kg) | 0.19 (NA) — Geometric CV was not calculated as data were available for only two participants. | 0.21 (NA) — Geometric CV was not calculated as data were available for only two participants. | 0.21 (26.6) | 0.22 (22.8) | 0.20 (54.9) | 0.21 (25.3) | 0.22 (25.9) | 0.23 (26.2) | 0.22 (12.9) | 0.20 (24.6) | 0.19 (27.5) | 0.22 (7.8) | NA (NA) — Geometric mean and CV were not calculated as data were available for only one participant.

10. Secondary Outcome: Terminal Half-Life (t½) of Selinexor
Description: t½ was, calculated as ln(2)/kel, where kel is elimination rate constant, calculated using linear regression on the terminal portion of the log-linear concentration versus time curve.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 4, 8, 24 and 48 hours post-dose on Day 1, 8 of Cycle 1 and Days 15, 16 or 17 of Cycle 2
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Selinexor (3 mg/m^2) | Selinexor (6 mg/m^2) | Selinexor (12 mg/m^2) | Selinexor (16.8 mg/m^2) | Selinexor (23 mg/m^2) | Selinexor (30 mg/m^2) | Selinexor (35 mg/m^2) | Selinexor (40 mg/m^2) | Selinexor (46 mg/m^2) | Selinexor (55 mg/m^2) | Selinexor (60 mg/m^2) | Selinexor (70 mg/m^2) | Selinexor (80 mg/m^2)
Number analyzed (Participants) | 2 | 2 | 6 | 12 | 12 | 21 | 13 | 8 | 9 | 7 | 3 | 4 | 1
hour | NA [5.5 to 6.1] — Median value was not calculated due to insufficient PK samples required for calculation. | NA [4.4 to 5.1] — Median value was not calculated due to insufficient PK samples required for calculation. | 6.2 [4.2 to 7.8] | 6.1 [3.1 to 8.7] | 6.9 [3.5 to 12.0] | 5.8 [3.9 to 8.4] | 6.2 [4.6 to 10.4] | 4.8 [2.7 to 9.8] | 5.7 [4.1 to 6.8] | 6.6 [5.4 to 10.1] | 5.9 [4.3 to 5.9] | 5.2 [5.0 to 6.0] | NA [5.5 to 5.5] — Median value was not calculated due to insufficient PK samples required for calculation.

11. Secondary Outcome: Number of Participants With Overall Response of Selinexor
Description: Objective response for each malignancy was defined using the disease response criteria by malignancy; For NHL (including DLBCL, PTCL, and CTCL), objective response included complete response (CR) and partial response (PR). For MM, objective response included stringent complete response (sCR), CR, very good partial response (VGPR), and PR. For WM, objective response included CR, VGPR, and PR. For CLL, ALL, and AML, objective response included complete remission and Partial remission. For CML, objective response includes complete cytogenic response, and complete hematologic response (CHR).
Time Frame: From first dose of study drug administration to end of treatment (up to 27 months)
Population: Efficacy analysis included all participants registered to the study who had either completed 1 cycle of treatment or discontinued treatment prior to completing the first cycle due to documented disease progression, death related to disease, or treatment-related toxicity.
Measure: Number; unit: participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Non-Hodgkin Lymphoma (NHL) Excluding DLBCL | Multiple Myeloma (MM) | Acute Myeloid Leukemia (AML) | Other Hematological Malignancies (ALL, CML and CLL)
Number analyzed (Participants) | 58 | 27 | 81 | 95 | 24
participants
  Complete response | 5 | 1 | 0 | 0 | 0
  Partial response | 7 | 8 | 6 | 0 | 0
  Morphologic complete remission | 0 | 0 | 0 | 4 | 0
  Partial remission | 0 | 0 | 0 | 3 | 1
  Complete cytogenetic response | 0 | 0 | 0 | 0 | 0
  Complete hematological response | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the first occurrence of objective response to first documented evidence of disease recurrence or progression. Participants without evidence of progression were censored at time of last evaluable disease assessment. Objective response was defined as any response of partial response/remission or better for all malignancies; for AML, a response of morphologic leukemia-free state is also included for ORR. Duration of response was calculated by Kaplan-Meier method.
Time Frame: From first dose of study drug administration to end of treatment (up to 27 months)
Population: Efficacy analysis included all participants who had either completed 1 cycle of treatment or discontinued treatment prior to completing the first cycle due to documented disease progression, death related to disease, or treatment-related toxicity. Here 'Overall Number of Participants Analyzed' signifies number of participants analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Non-Hodgkin Lymphoma (NHL) Excluding DLBCL | Multiple Myeloma (MM) | Acute Myeloid Leukemia (AML) | Other Hematological Malignancies (ALL, CML and CLL)
Number analyzed (Participants) | 12 | 9 | 7 | 11 | 1
Days | 335.5 [48 to NA] — Upper limit of 95% Confidence Interval (CI) was not estimable due to less than 50% death events. | 251 [36 to NA] — Upper limit of 95% CI was not estimable due to less than 50% death events. | 180 [57 to NA] — Upper limit of 95% CI was not estimable due to less than 50% death events. | 76 [29 to NA] — Upper limit of 95% CI was not estimable due to less than 50% death events. | NA [NA to NA] — Median and limits of 95% CI were not estimable due to less than 50% death events.

13. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was calculated from the date of first dose of study drug to first documented evidence of disease recurrence or progression or death due to any cause. Participants who were last known to be alive and without evidence of progression were censored at time of last evaluable disease assessment. If date of progression or death occurred after more than 1 missed disease assessment interval, participants were censored at the time of last evaluable disease assessment prior to the missed assessment.
Time Frame: Cycle 1 Day 1 to End of Treatment (up to 27 months)
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Non-Hodgkin Lymphoma (NHL) Excluding DLBCL | Multiple Myeloma (MM) | Acute Myeloid Leukemia (AML) | Other Hematological Malignancies (ALL, CML and CLL)
Number analyzed (Participants) | 58 | 27 | 81 | 95 | 24
Days | 47 [31 to 56] | 110 [28 to 274] | 57 [36 to 88] | 44 [36 to 52] | 57 [24 to 222]

14. Secondary Outcome: Duration of at Least Stable Disease
Description: Duration of at least stable disease was defined as the time from the date of first dose of study drug to first documented evidence of disease recurrence or progression. Participants without evidence of progression were censored at time of last evaluable disease assessment.
Time Frame: Cycle 1 Day 1 to End of Treatment (up to 27 months)
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Non-Hodgkin Lymphoma (NHL) Excluding DLBCL | Multiple Myeloma (MM) | Acute Myeloid Leukemia (AML) | Other Hematological Malignancies (ALL, CML and CLL)
Number analyzed (Participants) | 58 | 27 | 81 | 95 | 24
Days | 52 [32 to 79] | 114 [43 to 415] | 57 [43 to 100] | 80 [52 to 101] | 64 [21 to 283]

15. Secondary Outcome: Overall Survival
Description: Overall Survival was calculated from the date of first dose of study drug to date of death due to any cause. Participants who were last known to be alive were censored at time of last contact. Overall survival was calculated by Kaplan-Meier method.
Time Frame: Cycle 1 Day 1 to End of Treatment (up to 27 months)
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Non-Hodgkin Lymphoma (NHL) Excluding DLBCL | Multiple Myeloma (MM) | Acute Myeloid Leukemia (AML) | Other Hematological Malignancies (ALL, CML and CLL)
Number analyzed (Participants) | 58 | 27 | 81 | 95 | 24
Days | 138 [85 to NA] — Upper limit of 95% CI was not estimable due to less than 50% death events. | 423 [423 to NA] — Upper limit of 95% CI was not estimable due to less than 50% death events. | 366 [126 to NA] — Upper limit of 95% CI was not estimable due to less than 50% death events. | 76 [48 to 114] | 82 [50 to NA] — Upper limit of 95% CI was not estimable due to less than 50% death events.

ADVERSE EVENTS:
Time Frame: From first dose of study drug administration to end of treatment (up to 27 months)
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Non-Hodgkin Lymphoma (NHL) Excluding DLBCL | Multiple Myeloma (MM) | Acute Myeloid Leukemia (AML) | Other Hematological Malignancies (ALL, CML and CLL)
Serious Adverse Events (participants affected / at risk) | 33/58 | 7/27 | 52/81 | 73/95 | 13/24
Other Adverse Events (participants affected / at risk) | 58/58 | 27/27 | 80/81 | 94/95 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Large B-cell Lymphoma (DLBCL) (N=58) | Non-Hodgkin Lymphoma (NHL) Excluding DLBCL (N=27) | Multiple Myeloma (MM) (N=81) | Acute Myeloid Leukemia (AML) (N=95) | Other Hematological Malignancies (ALL, CML and CLL) (N=24)
Embolism (Vascular disorders) | 2 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 1 | 0 | 2 | 1 | 0
Small intestinal resection (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 4 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 5 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 6 | 0
Death (General disorders) | 1 | 0 | 0 | 3 | 1
Asthenia (General disorders) | 1 | 0 | 2 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 2 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 1 | 0
Unevaluable event (General disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (General disorders) | 3 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 6 | 12 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 1 | 0
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Leukostasis syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Central nervous system haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Encephalitis toxic (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 4 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 3 | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Headache (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 8 | 10 | 2
Sepsis (Infections and infestations) | 3 | 1 | 2 | 14 | 0
Lung infection (Infections and infestations) | 2 | 1 | 1 | 4 | 2
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 4 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 2 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Mucormycosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Diffuse Large B-cell Lymphoma (DLBCL) (N=58) | Non-Hodgkin Lymphoma (NHL) Excluding DLBCL (N=27) | Multiple Myeloma (MM) (N=81) | Acute Myeloid Leukemia (AML) (N=95) | Other Hematological Malignancies (ALL, CML and CLL) (N=24)
Hypotension (Vascular disorders) | 7 | 5 | 9 | 19 | 2
Hypertension (Vascular disorders) | 5 | 2 | 1 | 9 | 3
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 0 | 5 | 0
Hot flush (Vascular disorders) | 1 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 39 | 13 | 62 | 67 | 16
Pyrexia (General disorders) | 21 | 4 | 22 | 20 | 1
Oedema peripheral (General disorders) | 13 | 2 | 8 | 21 | 2
Asthenia (General disorders) | 2 | 4 | 14 | 7 | 0
Chills (General disorders) | 4 | 5 | 7 | 7 | 2
Gait disturbance (General disorders) | 6 | 1 | 7 | 2 | 2
Malaise (General disorders) | 5 | 2 | 5 | 2 | 1
Non-cardiac chest pain (General disorders) | 2 | 1 | 8 | 4 | 0
Oedema (General disorders) | 2 | 0 | 1 | 5 | 1
Peripheral swelling (General disorders) | 4 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 8 | 8 | 15 | 15 | 2
Insomnia (Psychiatric disorders) | 8 | 4 | 8 | 9 | 2
Anxiety (Psychiatric disorders) | 7 | 0 | 4 | 7 | 0
Depression (Psychiatric disorders) | 3 | 2 | 6 | 4 | 1
Agitation (Psychiatric disorders) | 5 | 0 | 6 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 2 | 8 | 8 | 4
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 6 | 5 | 4
Weight decreased (Investigations) | 14 | 10 | 32 | 31 | 3
Alanine aminotransferase increased (Investigations) | 7 | 2 | 8 | 10 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 1 | 7 | 10 | 2
Electrocardiogram QT prolonged (Investigations) | 2 | 1 | 3 | 10 | 5
International normalised ratio increased (Investigations) | 0 | 0 | 3 | 7 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 4 | 3 | 2
Sinus tachycardia (Cardiac disorders) | 4 | 0 | 1 | 3 | 0
Palpitations (Cardiac disorders) | 2 | 2 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 8 | 20 | 32 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 6 | 18 | 15 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 16 | 23 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 1 | 6 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 6 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 5 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 39 | 15 | 52 | 47 | 17
Anaemia (Blood and lymphatic system disorders) | 34 | 14 | 42 | 46 | 16
Neutropenia (Blood and lymphatic system disorders) | 23 | 12 | 31 | 23 | 10
Leukopenia (Blood and lymphatic system disorders) | 11 | 5 | 11 | 15 | 8
Lymphopenia (Blood and lymphatic system disorders) | 6 | 2 | 7 | 7 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 13 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 9 | 3
Dysgeusia (Nervous system disorders) | 13 | 6 | 16 | 22 | 1
Dizziness (Nervous system disorders) | 14 | 5 | 13 | 20 | 5
Headache (Nervous system disorders) | 7 | 4 | 11 | 16 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2 | 4 | 2 | 4
Neuropathy peripheral (Nervous system disorders) | 6 | 2 | 2 | 3 | 0
Syncope (Nervous system disorders) | 2 | 2 | 5 | 3 | 0
Amnesia (Nervous system disorders) | 1 | 2 | 1 | 3 | 0
Balance disorder (Nervous system disorders) | 3 | 2 | 2 | 0 | 0
Dysarthria (Nervous system disorders) | 3 | 1 | 0 | 1 | 0
Vision blurred (Eye disorders) | 15 | 4 | 21 | 21 | 6
Cataract (Eye disorders) | 2 | 2 | 6 | 3 | 1
Visual impairment (Eye disorders) | 5 | 1 | 3 | 1 | 0
Photopsia (Eye disorders) | 2 | 0 | 5 | 0 | 2
Dry eye (Eye disorders) | 2 | 2 | 1 | 2 | 0
Eye pain (Eye disorders) | 0 | 3 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 3 | 1 | 2 | 3 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1 | 5 | 0
Nausea (Gastrointestinal disorders) | 38 | 18 | 64 | 55 | 18
Vomiting (Gastrointestinal disorders) | 25 | 11 | 40 | 39 | 9
Diarrhoea (Gastrointestinal disorders) | 24 | 9 | 32 | 46 | 10
Constipation (Gastrointestinal disorders) | 15 | 9 | 15 | 29 | 6
Abdominal pain (Gastrointestinal disorders) | 11 | 3 | 9 | 10 | 4
Dyspepsia (Gastrointestinal disorders) | 8 | 2 | 9 | 5 | 1
Stomatitis (Gastrointestinal disorders) | 4 | 1 | 1 | 17 | 2
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 5 | 5 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 3 | 6 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 1 | 3 | 5 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 6 | 0
Haematuria (Renal and urinary disorders) | 3 | 1 | 5 | 6 | 3
Proteinuria (Renal and urinary disorders) | 3 | 2 | 4 | 3 | 4
Urinary incontinence (Renal and urinary disorders) | 1 | 3 | 2 | 2 | 2
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 2 | 5 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 4 | 2
Urinary retention (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 4 | 4 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 2 | 6 | 5 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3 | 7 | 2 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 8 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 5 | 6 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 2 | 19 | 13 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 4 | 13 | 15 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 7 | 14 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 6 | 6 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 5 | 6 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1 | 6 | 4 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 5 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 34 | 16 | 54 | 62 | 13
Hyponatraemia (Metabolism and nutrition disorders) | 25 | 7 | 36 | 34 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 5 | 12 | 22 | 2
Dehydration (Metabolism and nutrition disorders) | 7 | 4 | 27 | 15 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 10 | 0 | 23 | 18 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 4 | 6 | 19 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 7 | 6 | 18 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 6 | 7 | 18 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 4 | 6 | 13 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 3 | 3 | 11 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 4 | 5 | 9 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 | 1 | 1 | 10 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 5 | 0 | 3 | 6 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 2 | 0 | 6 | 5 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1 | 2
Urinary tract infection (Infections and infestations) | 5 | 3 | 7 | 5 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 9 | 4 | 1
Lung infection (Infections and infestations) | 5 | 2 | 3 | 3 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 4 | 9 | 1
Oral infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes